CLINICAL TRIAL: NCT06863948
Title: Pilot Randomized Controlled Trial of an Integrative Group Psychotherapy (Terebenin's Method) in Adults With Subclinical and Mild/Moderate Anxiety and Depression
Brief Title: Integrative Group Psychotherapy (Terebenin's Method) in Adults With Subclinical and Mild/Moderate Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SW023
Record Dates: First submitted 2025-02-20; First posted 2025-03-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Depression - Major Depressive Disorder
Keywords: deprssion; anxiety; psychotherapy; cortisol
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: "Terebenin's Method" (Experimental)
  Interventions: Other: Teribenin method
- Control Interventions (Active Comparator)
  Interventions: Other: Control Interventions

INTERVENTIONS:
Other: Teribenin method — Intervention: "Terebenin's Method"
  * Format:
  * Duration: 8 weeks, 1 session/week (2-3 hours).
  * Group size: 8-12 participants + 1-2 facilitators.
  * Structure of Each Session:
  * Introduction (10-15 min): Check-in, brief emotional reflection.
  * Main Phase (90-120 min): Psychodrama-like enactments, systemic constellation exercises, body-oriented practices, directive interpretation by the therapist.
  * Conclusion (15-20 min): Group reflection, integration, feedback.
  * Quality Assurance:
  * Audio/video recording (with consent) for supervision.
  * A standard protocol/manual specifying core techniques
  Arms: Intervention: "Terebenin's Method"
Other: Control Interventions — 1. Active Control (Preferred):
  * Group psychotherapy (CBT, Gestalt, or another recognized approach) matching the same 8-week schedule. 2. Waitlist Control (If Active Control Unavailable):
  * Participants receive no active intervention during the 8 weeks, then are offered therapy afterward (if applicable)
  Arms: Control Interventions

SUMMARY:
Title Pilot Randomized Controlled Trial of an Integrative Group Psychotherapy (Terebenin's Method) in Adults with Subclinical and Mild/Moderate Anxiety and Depression

Summary and Detailed Description (Single Text Block) Anxiety and depression are significant public health concerns, with the World Health Organization (WHO) estimating that depression affects over 280 million people worldwide. Anxiety disorders frequently co-occur with depression, creating additional burdens on individuals and society. Integrative psychotherapeutic approaches-which combine elements from psychodrama, family systemic methods, Gestalt therapy, and body-oriented techniques-have shown efficacy in mild to moderate depression, often matching or exceeding outcomes of single-orientation therapies.

Terebenin's Method is an integrative group psychotherapy that actively uses psychodrama-based enactments, systemic constellation exercises, body-oriented practices, and a directive therapeutic style, aiming to help participants gain insight into maladaptive or unconscious patterns and reduce anxiety and depressive symptoms. To objectively measure the impact of this intervention, salivary cortisol (a marker of hypothalamic-pituitary-adrenal axis activity) and salivary alpha-amylase (reflecting sympathetic nervous system activation) will be assessed. These biomarkers can help validate reported symptom improvements by capturing shifts in stress reactivity.

This pilot trial adopts a randomized (1:1), controlled, prospective design, enrolling 60 adults aged 18-60 with mild, moderate, or subclinical anxiety/depressive symptoms. Participants will be randomized to one of two arms: an 8-week Terebenin's Method group (1 session/week, 2-3 hours per session) or a control group that either receives a standard form of psychotherapy (active control) or is waitlisted (if an active control is not feasible). Assessors who administer rating scales or process saliva samples will remain blinded to group assignments.

Inclusion criteria include the ability to attend weekly sessions and adhere to saliva sampling procedures, with stable or no psychotropic medication use. Individuals with severe psychiatric disorders, acute suicidal risk, or other confounding factors (e.g., significant substance use, concurrent ongoing psychotherapy) will be excluded. Because this is a pilot study, each arm will have 30 participants (total n=60), providing initial data on feasibility, effect sizes, and biomarker changes.

Primary outcomes-depression (BDI-II or HAM-D) and anxiety (STAI or HADS-A)-will be assessed at baseline (T0), post-intervention (T1, ~8 weeks), and follow-up (T2, ~1-3 months). Secondary outcomes include quality of life (WHOQOL-BREF or SF-36), perceived stress (PSS), and therapeutic alliance (WAI). Salivary cortisol and alpha-amylase will be collected at three time points across two consecutive days (upon awakening, 30 minutes after awakening, and in the evening) at T0, T1, and T2. Analyses will focus on the cortisol awakening response (CAR) and area under the curve (AUC) for both biomarkers.

Data will be managed in a secure database with unique participant IDs. A repeated-measures ANOVA or mixed-effects model will be used to analyze changes in clinical and biomarker data from baseline to follow-up between the two groups. If normality assumptions are violated, nonparametric methods may be employed. Missing data will be handled by intent-to-treat principles (e.g., multiple imputation or last observation carried forward).

Overall, this pilot trial aims to: (1) demonstrate whether Terebenin's Method leads to greater reductions in anxiety and depressive symptoms compared to the control, (2) examine changes in objective stress biomarkers, and (3) refine the methodology and effect size estimates for a larger, fully powered randomized controlled trial.

DETAILED DESCRIPTION:
Anxiety and depression are among the most prevalent mental health disorders worldwide, often presenting with overlapping symptoms that amplify the burdens on affected individuals and healthcare systems. According to the World Health Organization (WHO), depression alone affects over 280 million people globally (approximately 3.5% of the population). Anxiety disorders share a similar high prevalence and frequently co-occur with depressive conditions. In response to these challenges, diverse psychotherapy modalities have emerged, including integrative approaches that combine principles from different schools (e.g., psychodrama, Gestalt, family systemic, and body-oriented methods) to enhance treatment effectiveness. Meta-analyses indicate that these integrative strategies can achieve effect sizes (Cohen's d) in the range of 0.60-0.90, making them viable-or in some cases superior-alternatives to single-orientation therapies for mild to moderate depression ].

Within this integrative framework, Terebenin's Method stands out as a structured group intervention designed to address subclinical, mild, or moderate anxiety and depression. Its core elements include psychodrama-inspired enactments (allowing participants to "act out" internal conflicts or emotional challenges in a safe group context), systemic constellation techniques (focusing on relational and family-system dynamics through phenomenological exploration), body-oriented practices (emphasizing awareness of somatic tension and facilitating emotional expression), and a directive therapeutic style (where the therapist actively interprets and guides group processes) . The method posits that enacting and witnessing others' enactments of unconscious or maladaptive patterns facilitates emotional insight and symptom reduction, concurrently reinforcing self-esteem, resilience, and a sense of control.

Besides patient-reported outcomes, growing attention has turned to physiological markers that can provide objective evidence of treatment efficacy. Salivary cortisol (CORT) is widely recognized as an indicator of hypothalamic-pituitary-adrenal (HPA) axis function, known to rise under chronic stress, depressive episodes, and anxiety conditions. Likewise, salivary alpha-amylase (sAA) reflects sympathetic nervous system (SNS) activation and tends to increase during acute stress. Research suggests that effective psychotherapies can lower or normalize these biomarkers, thereby validating clinical improvements captured through self-report and observer-rated scales.

Against this background, the present study is designed as a pilot randomized controlled trial (1:1 allocation) to evaluate the effects of Terebenin's Method in individuals aged 18-60 who exhibit subclinical to moderate anxiety or depressive symptoms. The study will enroll approximately 60 participants (30 per group), enabling the collection of feasibility data and effect size estimates to inform a larger, fully powered RCT. Participants will be randomly assigned to one of two arms: (1) an 8-week course of integrative group therapy using Terebenin's Method (weekly sessions of 2-3 hours, led by 1-2 trained facilitators with a group size of 8-12), or (2) a control condition that may consist of an active psychotherapeutic intervention (e.g., short-term cognitive-behavioral therapy or Gestalt group) conducted on a similar 8-week schedule, or a waitlist if the active control is not feasible.

Inclusion criteria require stable or no psychotropic medication use, absence of severe psychiatric disorders or acute suicidal risk, the ability to attend weekly sessions, compliance with saliva sampling, and written informed consent. Exclusion criteria encompass severe somatic illnesses preventing participation, current psychotherapy likely to confound results, and active substance use disorders unless in stable remission for more than six months.

Outcome measures will be collected at baseline (T0), post-intervention (~8 weeks, T1), and at follow-up (~1-3 months, T2). Primary clinical outcomes include depression scores (Beck Depression Inventory-II [BDI-II] or Hamilton Depression Rating Scale [HAM-D], administered by blinded evaluators) and anxiety scores (State-Trait Anxiety Inventory [STAI] or the anxiety subscale of the Hospital Anxiety and Depression Scale [HADS-A]). Secondary outcomes include quality of life (WHOQOL-BREF or SF-36), perceived stress (Perceived Stress Scale [PSS]), and therapeutic alliance (Working Alliance Inventory [WAI]). Physiological outcomes center on salivary cortisol and alpha-amylase, sampled three times a day (upon awakening, 30 minutes post-awakening, and in the evening) over two consecutive days at T0, T1, and T2. Key metrics will be the cortisol awakening response (CAR) and area under the curve (AUC) for both biomarkers.

Data management involves the use of standardized collection kits (e.g., Salivette®) and secure databases with unique participant IDs. Statistical analysis will follow an intent-to-treat approach, with repeated-measures ANOVA or mixed-effects models used to compare within- and between-group changes over time for both clinical and biomarker data. Normality violations may prompt nonparametric alternatives. Missing data will be handled via multiple imputation or last observation carried forward. A two-tailed alpha of p < 0.05 will be the threshold for statistical significance.

In summary, this pilot trial seeks to evaluate whether Terebenin's Method, an integrative group psychotherapy approach, yields clinically meaningful improvements in anxiety and depression while concurrently influencing objective biological markers of stress (salivary cortisol and alpha-amylase). The study's results will guide refinement of the intervention protocol, confirm or adjust effect size estimates, and lay the groundwork for a more extensive randomized controlled trial to rigorously test Terebenin's Method in larger and more diverse populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60.

  * Subclinical, mild, or moderate anxiety/depressive symptoms (screened via HADS, BDI-II, STAI).
  * No current psychotropic medication use or on a stable dose for ≥4 weeks with no planned changes.
  * Ability to attend weekly group sessions for 8 weeks + follow-up visits, including saliva sample collection.
  * Provision of written informed consent.

Exclusion Criteria:

* Severe psychiatric disorders (e.g., schizophrenia, bipolar disorder in a manic phase, major depression with psychotic features).

  * Significant suicidal risk requiring urgent intervention.
  * Severe somatic illness impeding participation.
  * Active substance use disorder unless in stable remission for >6 months.
  * Ongoing psychotherapy that could confound results.
  * Inability to comply with saliva collection (e.g., shift work, severe sleep disturbances).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-10-12 (Actual)

PRIMARY OUTCOMES:
Depression Scores | 3 months
  The Beck Depression Inventory-II is a 21-item self-report scale measuring the severity of depressive symptoms. Each item is scored from 0 to 3, with total scores ranging from 0 (no depression) to 63 (severe depression). Higher scores indicate a worse outcome .
Anxiety Score | 3 months
  The State-Trait Anxiety Inventory contains two 20-item subscales assessing state anxiety and trait anxiety. Each item is scored from 1 to 4, leading to subscale scores ranging from 20 to 80. Higher scores indicate a worse outcome (i.e., higher levels of anxiety).

SECONDARY OUTCOMES:
Quality of Life / Well-Being | 3 months
  The World Health Organization Quality of Life-BREF( WHOQOL-BREF) is a 26-item measure assessing four domains (physical health, psychological health, social relationships, and environment). Scores in each domain can range from 0 to 100.
Perceived Stress | 3 months
  The Perceived Stress Scale (PSS) is a 10-item self-report questionnaire measuring the degree to which situations in one's life are appraised as stressful. Total scores range from 0 to 40.
Therapeutic Alliance | 3 months
  The Working Alliance Inventory (WAI) measures the therapeutic alliance between a clinician and client. In its short form (WAI-SF), there are 12 items rated on a 7-point scale, giving total scores ranging from 12 to 84.
Salivary Cortisol (CORT): | 3 months
  Sampling: 3 times a day (upon awakening [C0], 30 min after awakening [C0+30], and evening)
Salivary Alpha-Amylase | 3 months
  Collected at the same times as cortisol.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Technologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No